CLINICAL TRIAL: NCT05497245
Title: Development of Mobile Application Based Breastfeeding Education Program and Evaluation of the Program Effectiveness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, ZEHRA ACAR, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 121S326
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Breastfeeding, Exclusive
Keywords: breastfeeding; breastmilk; mobile health
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): mobile app-based breastfeeding education
  Interventions: Other: mobile app-based breastfeeding education
- control group (No Intervention): rutin health care

INTERVENTIONS:
Other: mobile app-based breastfeeding education — The main screen of the application used to be six screens. These six screens; Breastfeeding, Expressing, Contingencies, Frequently asked questions and my Breastfeeding Log and Breastfeeding diary. Mothers could record the number and duration of breastfeeding, milking status, the baby's height and weight, if it was a measure, the breastfeeding problem and solutions they encountered, on the "Breastfeeding Introduction" tab, and they could follow their breastfeeding status in the "Breastfeeding Diary" tab.
  Arms: intervention group

SUMMARY:
Purpose of Research: The purpose of this research is to develop and evaluate the effectiveness of a mobile application-based breastfeeding education program.

Research Hypotheses H1: Exclusive breastfeeding rate is higher for mothers in the experimental group than the mothers in the control group in the fourth postpartum week.

H2: The mothers in the experimental group had higher scores on the Evaluation of Breastfeeding Problems in the fourth week after delivery than the mothers in the control group.

H3: Exclusive breastfeeding rate is higher for the mothers in the experimental group than the mothers in the control group in the eighth postpartum week.

H4: The mothers in the experimental group had higher scores on the Evaluation of Breastfeeding Problems at the eighth postpartum week than the mothers in the control group.

In the first stage of the research, a mobile application-based breastfeeding education program was developed and piloted. In the second stage of the study, the mobile application-based breastfeeding education program was applied to the primiparous mothers in the experimental group for eight weeks, starting from the first day of postpartum.The control group received only routine health care.

617 / 5.000 Çeviri sonuçları Personal Information Form, Breastfeeding Evaluation Scale and Breastfeeding Problems Evaluation Scale were applied to the mothers in the Experimental and Control groups on the first postpartum day.

* A mobile application was installed on the phones of the mothers in the experimental group and information was provided. The control group benefited only from routine nursing care.
* Infants' Physical Development Monitoring Form, Breastfeeding Monitoring Form, Breastfeeding Problems Evaluation Scale will be applied to the mothers in the experimental and control groups in the fourth and eighth weeks postpartum.
* Mobile Application Evaluation Form was also applied to the experimental group in the eighth week.

DETAILED DESCRIPTION:
The research consists of two stages. In the first stage, the mobile application was developed and a pilot application was made with 6 mothers in the testing of the application. For the second stage of the research, all primiparous mothers in Istanbul University Cerrahpaşa Medical Faculty Hospital between September 2021 and August 2022 constituted the population of the research. The sample of the study consisted of primiparous mothers who met the inclusion criteria and volunteered to participate in the study. The sample of the study formed the Experiment and Control group. Primiparous mothers in the experimental group were included in the mobile application-based breastfeeding education program, and the primiparous mothers in the control group were not included in this program and only benefited from the hospital's routine care services (Figure 1.) Power analysis was performed using the G-Power program to determine the number of samples. According to Cohen's effect size coefficients; According to the calculation made by assuming that the evaluations to be made between two independent groups will have a large effect size (d=0.8), when α: 0.05 and 90% power are taken, there should be at least 34 people for each group, considering the losses that may occur during the research process. A total of 80 primiparous mothers, 40 for one group, were planned to be included in the study..

The research consists of two stages. The first stage of the research consists of creating the information content of the mobile application-based breastfeeding education program, developing the application and making the pilot application. In the second stage of the study, primiparous mothers in the experimental group were included in the mobile application-based breastfeeding education program, while the mothers in the control group were not included in any practice other than routine nursing care. Data from mothers in the experimental and control groups were collected on postpartum first day, fourth week, and eighth week.

The first stage of the research Creating the content of the mobile application-based breastfeeding program In the first stage of the research, the content of the mobile application-based breastfeeding program was prepared in line with the literature. Presenting the content of the program on a scientific basis and the measurement and evaluation of education/programs in the world are now stated as an important criterion of evidence-based studies. For this reason, the content of the application was prepared with reference to the current sources of "World Health Organization" and "Ministry of Health". After the content was prepared, the development process of the mobile application was started.

Development of a mobile application-based breastfeeding program The development of the mobile application consists of six main stages: design, development, testing, reporting, maintenance and deployment. Design phase; It consists of evaluating the requirements analysis, considering the User Interface (UI) and user experience (UX) standards, printing the design as Mock-Up and submitting it for approval, and revising it in line with the data notifications. Development phase; development in line with the approved design, interaction via cloud (Cloud) service (Firebase), and development of the application on Cross-Platform as IOS and Android. Development phase; development in line with the approved design, interaction via cloud (Cloud) service (Firebase), and development of the application on Cross-Platform as IOS and Android. Development phase; development in line with the approved design, interaction via cloud (Cloud) service (Firebase), and development of the application on Cross-Platform as IOS and Android. Test phase; It consists of preparing the pilot-test environment, producing the IPA for the IOS version, producing the APK file for Android and conducting development tests. Reporting phase; consists of reporting and sharing the information received from the user. Maintenance phase; In the testing process, it consists of the process of making adjustments and improvements in the application in line with the feedback. The last stage, the distribution stage, is; It consists of obtaining certificates for Android and Apple, preparing necessary images for Android and Apple market environment, obtaining distribution approval by Apple and Android and uploading them to Apple and Android Market. In this direction, first of all, a special logo was designed for the application. Afterwards, the prepared content was integrated into the application. By clicking on the sign up tab at the first login of the application, an e-mail and password were created and the login application was registered, and the next login was made automatically. The information page of the application contained brief information about the application and three pages on the importance of breastfeeding and breast milk. Afterwards, information about the mother's name, baby's name, baby's gender and baby's birth weight was filled and the application was entered. These two screens were reserved for the first entry only. The main screen of the application used to be six screens. These six screens; Breastfeeding, Expressing, Contingencies, Frequently asked questions and my Breastfeeding Log and Breastfeeding diary. Mothers could record the number and duration of breastfeeding, milking status, the baby's height and weight, if it was a measure, the breastfeeding problem and solutions they encountered, on the "Breastfeeding Introduction" tab, and they could follow their breastfeeding status in the "Breastfeeding Diary" tab. In addition, notifications were sent once at the first entry to the application, and then 2-3 times a week to increase the breastfeeding motivation of the mothers.

The notification sent on the first login to the application; "Dear mom, your breastfeeding journey has begun. In this process, you can access the information you need through the application, keep a diary at the breastfeeding entrance and follow the breastfeeding process…"

Making a pilot application With the development of the application, the pilot application was started. Six mothers who met the inclusion criteria were included. The link of the application was sent to Android-operated phones via google drive in order to prevent sharing, and application invitation mail was sent to IOS-operated phones, application registrations were made through the app store, and the application was accessed by entering the code via the "Test Flight" application.

Mothers expressed the progress error on the breastfeeding home page, this technical issue was edited by the mobile application developer. In addition, mothers stated that they can have videos in the application and that receiving notifications will ensure the continuity of breastfeeding login. With these suggestions, the papers were systematized. No video is included in the application as it may negatively affect the usability of the application.

Second phase of the research In the second stage of the study, mothers who met the criteria for inclusion in the sampling were informed about the purpose, content and method of the study, and informed consent was obtained from the mothers who agreed to participate in the study. Following the CONSORT 2017 (Updated Guidelines for Reporting Randomized Parallel Group Studies) report, mothers were randomly assigned to the Experiment and Control groups using a simple random numbers table on https://www.random.org/integers/. Personal Information Form, Breastfeeding Evaluation Scale and Breastfeeding Problems Evaluation Scale were applied to the mothers in the Experimental and Control groups on the first postpartum day. The mobile application was installed on the phones of the mothers in the experimental group and they were informed about the content and use of the application. The control group benefited only from routine nursing care. Infants' Physical Development Monitoring Form, Breastfeeding Monitoring Form, Breastfeeding Problems Evaluation Scale were applied to the mothers in the experimental and control groups in the fourth and eighth weeks postpartum. The baby's weight, height and head circumference, which was included in the Baby's Physical Development Monitoring Form, was measured at the "Family Health Center". Due to the reduction of the difference between the measurements, the babies were asked to be weighed with clean diapers and without clothes. The mothers who had difficulty in filling out the questions online were contacted by the researcher and they were asked to read and answer the questions. In addition, the Mobile Application Evaluation Form was applied to the experimental group in the eighth week.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* Primiparous,
* Babies born at term (> 37 weeks of pregnancy or weight > 2500 g) and no health problems that prevent suckling
* Planning to breastfeed,
* Having a smart phone and effective usage skills,
* Mothers who agreed to participate in the study for eight weeks were included in the sample.

Exclusion Criteria:

* Being the first born,
* Having multiple pregnancy,
* Having a physical and/or mental health problem
* Having a risky newborn,
* Having a history of breast surgery or breast reduction. The puerperant women eligible for inclusion in the sampling were assigned to the experimental and control groups by randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
breastmilk exclusive | postpartum 1st day- postpartum 8th week
  rate of exclusive breastfeeding for eight weeks
breastfeeding problem | postpartum 1st day- postpartum 8th week
  rate of breastfeeding problem eight weeks
baby's physical development | postpartum 1st day- postpartum 8th week
  development of baby's weight, height and head circumference

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang CJ, Chaovalit P, Pongnumkul S. A Breastfeed-Promoting Mobile App Intervention: Usability and Usefulness Study. JMIR Mhealth Uhealth. 2018 Jan 26;6(1):e27. doi: 10.2196/mhealth.8337. PMID 29374000
- [Background] Ferraz Dos Santos L, Borges RF, de Azambuja DA. Telehealth and Breastfeeding: An Integrative Review. Telemed J E Health. 2020 Jul;26(7):837-846. doi: 10.1089/tmj.2019.0073. Epub 2019 Oct 18. PMID 31633467
- [Background] Doan TTD, Binns C, Pham NM, Zhao Y, Dinh TPH, Bui TTH, Tran TC, Nguyen XH, Giglia R, Xu F, Lee A. Improving Breastfeeding by Empowering Mothers in Vietnam: A Randomised Controlled Trial of a Mobile App. Int J Environ Res Public Health. 2020 Jul 31;17(15):5552. doi: 10.3390/ijerph17155552. PMID 32752026
- [Background] Schindler-Ruwisch JM, Roess A, Robert RC, Napolitano MA, Chiang S. Social Support for Breastfeeding in the Era of mHealth: A Content Analysis. J Hum Lact. 2018 Aug;34(3):543-555. doi: 10.1177/0890334418773302. Epub 2018 May 22. PMID 29787686